CLINICAL TRIAL: NCT05129410
Title: Clinical Study of MMF in Treatment of IIM-ILD and Its Effect on Peripheral Blood Treg Cells
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-194
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Inflammatory Myopathy; Interstitial Lung Disease
Keywords: Idiopathic inflammatory myopathy; interstitial lung disease; Mycophenolate Mofetil; Treg; Th17
MeSH Terms: conditions — Myositis; Lung Diseases, Interstitial | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: A single-arm open-label pilot observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A single-arm open-label pilot observational study (Experimental): Patients were received prednisone(0.5mg-1mg/kg/day) and a combination with MMF (1.5g-2.0g/d).
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 1. Prednisone 0.5-1.0 mg/kg/d, the dose was gradually reduced, and after 4 weeks, the dose was reduced by 5mg every two weeks, and then reduced to 10mg/d for 4-6 months after oral administration for 3 months, and then reduced to 7.5mg/d for maintenance therapy until 12 months;
  2. MMF1.5g-2.0g/d

SUMMARY:
Interstitial lung disease (ILD) is a common pulmonary manifestation of idiopathic inflammatory myopathy (IIM). The overall 5-year mortality is 50%. The prognosis is poor and the treatment is challenging.At present, according to the consensus of IIM-ILD experts, glucocorticoids as first-line treatment are often used in high doses and have a variety of adverse reactions. Previous studies have shown that cyclophosphamide (CYC) is effective for IIM-ILD and tends to be used in rapidly progressive interstitial lung disease（RP-ILD）or refractory ILD. However, CYC is an alkylating agent with many toxic and side effects. It is prone to gonadal inhibition, infection, tumor, hemorrhagic cystitis and other risks. At present, Mycophenolate mofetil (MMF) has been widly used in the treatment of IIM, systemic lupus erythematosus (SLE), ANCA associated vasculitis (AAV). The observational research on MMF in the treatment of IIM-ILD shows that it can delay the progress of pulmonary fibrosis and can be used as the first-line treatment of IIM-ILD. Moreover, immune tolerance caused by defects in the number and/or quality of regulatory T cells (Treg) is considered to be a key source of autoimmune diseases. However, it is unclear whether MMF can improve the immune status of IIM-ILD by increasing Treg cells. The aim of this study was to evaluate the effect of MMF for IIM-ILD and its effcts on Treg through a prospective open single arm study, and provide a theoretical basis for the individualized treatment of IIM-ILD, which has important clinical significance.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a common pulmonary manifestation of idiopathic inflammatory myopathy (IIM), with an incidence ranging from 23.1 to 65%. The treatment of IIM patients with ILD is challenging, and the overall 5-year mortality is 50%. The disease process of ILD from stable or slow to rapid. Increased mortality and poor prognosis were observed, which needs active treatment. At present, according to the consensus of IIM-ILD experts, glucocorticoids as first-line treatment are often used in high doses, but have a variety of adverse reactions. Previous studies have shown that cyclophosphamide (CYC) is effective for IIM-ILD and tends to be used in rapidly progressive interstitial lung disease（RP-ILD）or refractory ILD. However, CYC is an alkylating agent with many toxic and side effects. It is prone to gonadal inhibition, infection, tumor, hemorrhagic cystitis and other risks. Mycophenolate mofetil (MMF) has been widly used in the treatment of IIM, systemic lupus erythematosus (SLE), ANCA associated vasculitis (AAV). The observational research on MMF in the treatment of IIM-ILD shows that it can delay the progress of pulmonary fibrosis and can be used as the first-line treatment of IIM-ILD. Moreover, immune tolerance caused by defects in the number and / or quality of regulatory T cells (Treg) is considered to be a key source of autoimmune diseases. In transplant patients, studies have found that the combination of MMF and tacrolimus can increase the number of Treg cells in peripheral blood, suggesting that MMF has a certain regulatory effect on Treg cells. Therefore, it is unclear whether MMF can improve the immune status of IIM-ILD by increasing Treg cells, so as to improve the prognosis of the disease. However, it is unclear whether MMF can improve the immune status of IIM-ILD by increasing Treg cells. The aim of this study was to evaluate the effect of MMF for IIM-ILD and its effcts on Treg through a prospective open single arm study, and provide a theoretical basis for the individualized treatment of IIM-ILD.This was a single-arm open-label pilot observational study. Patients were received prednisone (0.5mg-1.0mg/kg/d ) combined with MMF(1.5g-2.0g/d) for 12 months, 4 weeks later, reduced 5mg every two weeks to 10mg/d orally for 3 months, gradually reduced to 7.5mg/ day until 12 months.

ELIGIBILITY:
Inclusion Criteria:

* meet the PM/DM diagnostic criteria according to Bohan-Peter
* consistent with ILD diagnosis
* predicted forced vital capacity (FVC) of at least 50%
* patients who did not use immunosuppress agents (including but not limited to cyclophosphamide, cyclosporine, leflunomide, azathioprine, tacrolimus, etc.) at the time of screening, or who had stopped taking drugs for ≥3 months.

Exclusion Criteria:

* Anti MDA5 antibody positive DM and necrotizing myopathy
* patients if they had other connective tissue diseases, an underlying cancer, a concomitant active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
FVC % predicted | 12 months
  Percentage of predicted FVC

SECONDARY OUTCOMES:
DLCO % predicted | 12 months
  Percentage of predicted DLCO
Lung high resolution CT score | 12 months
  Lung high resolution CT score
TDI | 12 months
  Transitional dyspnoea index
TIS | 12 months
  Clinical response
Overall survival rate | 12 months
  Overall survival rate%
Infection rate | 12 months
  Infection rate%

CONTACTS AND LOCATIONS:
Overall Officials: Lan He, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Department of Rheumatology,the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Long K, Danoff SK. Interstitial Lung Disease in Polymyositis and Dermatomyositis. Clin Chest Med. 2019 Sep;40(3):561-572. doi: 10.1016/j.ccm.2019.05.004. PMID 31376891
- [Result] Nihtyanova SI, Brough GM, Black CM, Denton CP. Mycophenolate mofetil in diffuse cutaneous systemic sclerosis--a retrospective analysis. Rheumatology (Oxford). 2007 Mar;46(3):442-5. doi: 10.1093/rheumatology/kel244. Epub 2006 Aug 9. PMID 16899504
- [Result] Edge JC, Outland JD, Dempsey JR, Callen JP. Mycophenolate mofetil as an effective corticosteroid-sparing therapy for recalcitrant dermatomyositis. Arch Dermatol. 2006 Jan;142(1):65-9. doi: 10.1001/archderm.142.1.65. PMID 16415388
- [Result] Antiga E, Kretz CC, Klembt R, Massi D, Ruland V, Stumpf C, Baroni G, Hartmann M, Hartschuh W, Volpi W, Del Bianco E, Enk A, Fabbri P, Krammer PH, Caproni M, Kuhn A. Characterization of regulatory T cells in patients with dermatomyositis. J Autoimmun. 2010 Dec;35(4):342-50. doi: 10.1016/j.jaut.2010.07.006. Epub 2010 Sep 16. PMID 20843660